CLINICAL TRIAL: NCT01678157
Title: Use of Strattice in the Laparoscopic Suture Closure of a Paraesophageal Hernia
Brief Title: Use of Strattice Mesh in Paraesophageal Hernia Surgery
Acronym: Strattice
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: LifeCell (Industry)
Responsible Party: Sponsor
Other Study IDs: 0314-11-FB
Record Dates: First submitted 2012-08-29; First posted 2012-09-03 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Hernia; Hernia, Esophageal; Hernia, Paraesophageal; Hiatal Hernia; Paraesophageal Hiatal Hernia; Sliding Esophageal Hernia; Sliding Hiatal Hernia
Keywords: Esophageal Hernia; Hernia, Esophageal; Hernia, Paraesophageal; Hiatal Hernia; Paraesophageal Hiatal Hernia; Sliding Esophageal Hernia; Sliding Hiatal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Documented symptomatic paraesophageal hernia: 1. Documented symptomatic paraesophageal hernia.
  2. Greater than 5 cm hiatal hernia on upper gastrointestinal study.
  3. Evidence that the stomach or other viscera is present in the hernia and does not spontaneously reduce from the mediastinum.
  4. Significant symptoms or signs of a paraesophageal hernia including but not limited to heartburn,dysphagia, chest pain, shortness of breath, postprandial abdominal pain, early satiety, odynophagia, or chronic anemia.
  5. Consenting adult 19 years of age or older
  6. Must be able to participate in follow-up evaluation.
  7. Free of cognitive impairment

SUMMARY:
The objective of this study is to examine the safety and efficacy of porcine acellular dermal matrix mesh (Strattice; LifeCell Corp., Branchburg, NJ) in crural reinforcement of laparoscopic large paraesophageal hernia repair.

DETAILED DESCRIPTION:
Prosthetic reinforcements reduce recurrence rates; the choice of optimal prosthetic, either synthetic or biosynthetic, for crural reinforcement is controversial. The objective of this study is to examine the safety and efficacy of porcine acellular dermal matrix mesh (Strattice; LifeCell Corp., Branchburg, NJ) in crural reinforcement of laparoscopic large paraesophageal hernia repair. Strattice is a commonly used mesh in hernia repair. 35 adult (>19 years of age) patients will be selected based on inclusion and exclusion criteria. Patients who meet the criteria will be enrolled in the study. Information related to recurrence rates based on follow-up visits will be analyzed to determine the efficacy of Strattice in the prevention of large hernia recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Documented symptomatic paraesophageal hernia.
* Greater than 5 cm hiatal hernia on upper gastrointestinal study.
* Evidence that the stomach or other viscera is present in the hernia and does not spontaneously reduce from the mediastinum.
* Significant symptoms or signs of a paraesophageal hernia including but not limited to heartburn, dysphagia, chest pain, shortness of breath, postprandial abdominal pain, early satiety, odynophagia, or chronic anemia.
* Consenting adult 19 years of age or older
* Must be able to participate in follow-up evaluation.
* Free of cognitive impairment

Exclusion Criteria:

* Children and adolescents (19 years of age or younger).
* Pregnant and breast feeding patients.
* Vulnerable subjects such as pregnant women, children less than 19 years age, and decisionally impaired persons.
* Patients with previous operation of the esophagus or stomach.
* Patients with associated gastrointestinal diseases that require extensive medical or surgical intervention that might interfere with quality of life assessment (e.g. Crohn's disease).
* Patients with emergent operation for acute gastric volvulus.
* Patients with known sensitivity to porcine material.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over 19 years of age with paraesophageal hernia greater than 5 cm.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-03-05 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence | 1 year post-surgery
  A barium swallow test with x-rays will be performed to assess recurrence of hernia, if any

SECONDARY OUTCOMES:
Recurrence of reflux symptoms | 2 weeks, 6 months and 1 year post-surgery
  Patients will be evaluated for recurrence of reflux symptoms at the three postoperative visits. If recurrence warrants, a barium swallow with x-rays will be performed prior to 1-year primary outcome barium swallow test

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Oleynikov, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States